CLINICAL TRIAL: NCT03654053
Title: Effect of Simvastatin on Hepatic Decompensation and Death in Subjects With High-risk Compensated Cirrhosis
Brief Title: Multi-Center Study of the Effects of Simvastatin on Hepatic Decompensation and Death in Subjects Presenting With High-Risk Compensated Cirrhosis
Acronym: SACRED
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GAST-010-19F; VOCAL-001 (Other: Department of Veterans Affairs)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis
Keywords: cirrhosis; hepatic decompensation; HMG-coA reductase; hepatocellular carcinoma; clinical trial; Human
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin (Experimental): Simvastatin 40mg PO once at bedtime for up to 24 months. Note: all enrolled subjects will trial 20mg once at bedtime for two weeks as lead-in to determine tolerability prior to randomization.
  Interventions: Drug: Simvastatin 40mg
- Placebo (Placebo Comparator): Placebo 40mg PO once at bedtime for up to 24 months. Note: all enrolled subjects will trial 20mg once at bedtime for two weeks as lead-in to determine tolerability prior to randomization.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo taken once nightly at bed time.
  Other Names: Placebo
  Arms: Placebo
Drug: Simvastatin 40mg — Simvastatin 40mg taken once nightly at bed time.
  Other Names: Simvastatin
  Arms: Simvastatin

SUMMARY:
This phase III, randomized, double-blind, placebo-controlled, multi-center study seeks to test whether simvastatin, a statin usually used to lower cholesterol to prevent heart problems and strokes, can lower the risk of hepatic decompensation (developing symptoms of cirrhosis) in U.S. Veterans who have compensated cirrhosis (the liver is scarred and damaged but there are no symptoms). The study will also explore how changes or differences in genes effect the safety and effectiveness of using statins and how the use of statins affects quality of life.

DETAILED DESCRIPTION:
HMG-coA reductase inhibitors (statins), independent of cholesterol-lowering effects, are beneficial in liver diseases by reducing endothelial dysfunction, intrahepatic vasoconstriction, inflammation and fibrosis, and can reduce portal vein blood pressure. Clinically significant portal hypertension (hepatic vein wedge pressure greater than or equal to 10mmHg) is the most important predictor of decompensation and death in patients with cirrhosis.

This randomized, double-blind, placebo-controlled, multi-center Phase III interventional study seeks to demonstrate that statin therapy in patients with cirrhosis at high-risk for hepatic decompensation will reduce the incidence of hepatic decompensation, hepatocellular carcinoma or all-cause mortality.

Patients with compensated cirrhosis at high-risk for hepatic decompensation will be stratified based on the presence or absence of varices and randomized to simvastatin 40mg/day for up to 24 months. Patients will be observed for the development of hepatic decompensation (variceal hemorrhage, ascites, encephalopathy), hepatocellular carcinoma, liver-related death, death from any cause, and/or complications of statin therapy. Additionally, the interaction of SLCO1B1 and KIF6 polymorphisms on safety and clinical efficacy of statin therapy and the impact of statin exposure on health-related quality of life in patients with compensated cirrhosis will be examined.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran
* Cirrhosis due to chronic viral hepatitis, or alcohol or non-alcoholic fatty liver
* Compensated cirrhosis (history of endoscopically-confirmed variceal hemorrhage, absence of overt ascites, history of overt non-precipitated encephalopathy)
* Age > 18 and <= 80
* High risk of cirrhosis decompensation as defined by any of the following:

  * Presence of esophageal varices on endoscopy
  * Presence of portosystemic collaterals on imaging as determined by a body radiologist
  * Fibroscan VCTE >= 20kPa
  * Platelet count <= 125 K/mm
  * 44 total points (~50% of clinically significant portal hypertension using the ANTICIPATE Nomogram)
* Competent to provide informed consent

Exclusion Criteria:

* Prior exposure to any statin within 6 months
* Prior allergy or sensitivity to simvastatin
* History of variceal hemorrhage confirmed endoscopically within the previous 3 years
* Presence of overt ascites or treatment with diuretics for ascites with 6 months
* History of chronic, recurrent or episodic overt hepatic encephalopathy with asterixis within 6 months
* History of hepatocellular carcinoma
* Child-Turcotte-Pugh C Stage (CTP Score > 9)
* Prior receipt of organ transplant
* Participation in another pharmacological clinical trial within 3 months of the current study
* Pregnancy or anticipated pregnancy within 2 years
* Breast Feeding
* Patients with life expectancy < 3 years due to comorbid conditions
* Independent indication for initiation of statin therapy
* Patients with any form of clinical atherosclerotic cardiovascular disease (ASCVD)
* Patients with primary LDL-C < 190 mg/dl
* Patients with diabetes mellitus, age 40-75 years, with LDL-C levels >=130 mg/dl
* Need for concomitant administration of potent inhibitors of CYP34A4 enzymes (medications or other supplements that should not be taken with simvastatin, including cyclosporine, danazol, gemfibrozil, fenofibrate, extended release niacin, itraconazole, ketoconazole, voriconazole, HIV protease inhibitors, boceprevir, telaprevir, macrolide antibiotics - erythromycin, clarithromycin, telithromycin, nefazadone, amlodipine, verapamil, diltiazem, dronedarone, amiodarone, renolazine, lomitapide, and cobicistat)
* Prior TIPSS shunt
* Hemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival free from hepatic decompensation | 24 months
  Occurrence of hepatic decompensation measured by first variceal hemorrhage, or development of ascites, or onset of hepatic encephalopathy, or hepatocellular carcinoma.

SECONDARY OUTCOMES:
Liver-related death | 24 months
  Occurrence of death after hepatic decompensation, or hepatocellular carcinoma or transplantation
Survival free from major cardiac events | 24 months
  Occurrence of acute myocardial infarction, or unstable angina, or acute ischemic stroke, or coronary revascularization.
Change in patient health-related quality of life | 12 months
  Clinically significant change in score from baseline to month 12 as assessed by the PROMIS-29 questionnaire
Statin-related hepatotoxicity | 24 months
  Occurrence of hepatotoxicity defined as Grade 3 liver toxicity per CTCAE 5.0 ( 5 times upper limit of normal as defined by local laboratory- transaminases)
Myositis | 24 months
  Occurrence of myositis defined as either Grade 3 myositis (pain associated with severe weakness; limiting self care Activities Daily Living {ADL}) OR Grade 4 creatine phosphokinase by CTCAE 5.0 ( 10x upper limit of normal)
Rhabdomyolysis | 24 months
  Occurrence of rhabdomyolysis defined as Grade 3 (symptomatic, urgent intervention indicated)
Hepatotoxicity | 24 months
  Liver enzyme testing (AST, ALT, alkaline phosphatase, total bilirubin) at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: David E. Kaplan, MD MSc, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (11):
- United States (11):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Robley Rex VA Medical Center, Louisville, KY, Louisville, Kentucky
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Brooklyn Campus of the VA NY Harbor Healthcare System, Brooklyn, NY, Brooklyn, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon request following completion of a DUA for purposes of verification and meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following closure of study database
Access Criteria: Data use / data transfer agreement

REFERENCES:
- [Background] Kaplan DE, Mehta R, Garcia-Tsao G, Albrecht J, Aytaman A, Baffy G, Bajaj J, Hernaez R, Hunt K, Ioannou G, Johnson K, Kanwal F, Lee TH, Monto A, Pandya P, Schaubel D, Taddei TH. SACRED: Effect of simvastatin on hepatic decompensation and death in subjects with high-risk compensated cirrhosis: Statins and Cirrhosis: Reducing Events of Decompensation. Contemp Clin Trials. 2021 May;104:106367. doi: 10.1016/j.cct.2021.106367. Epub 2021 Mar 24. PMID 33771685

DOCUMENTS (1):
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03654053/ICF_000.pdf